CLINICAL TRIAL: NCT04264000
Title: Platelet-rich Plasma Injection for Ulnar Neuropathy at Elbow: A Randomized Double-blind Trial
Brief Title: Platelet-rich Plasma Injection for Ulnar Neuropathy at Elbow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yung-Tsan Wu (Other)
Responsible Party: Sponsor-Investigator, Yung-Tsan Wu, Attending Physician and associated professor of Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Organization: Tri-Service General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRP for ulnar neuropathy
Record Dates: First submitted 2020-02-04; First posted 2020-02-11 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Ulnar Neuropathy at Elbow
Keywords: Ulnar Neuropathy at Elbow; platelet-rich plasma; Perineural injection
MeSH Terms: interventions — Glucose

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- platelet-rich plasma (Experimental): The perineural injection with PRP is a potential treatment for peripheral entrapment neuropathy
  Interventions: Drug: platelet-rich plasma
- 5% dextrose (Active Comparator): The perineural injection of 5% dextrose is a novel management for peripheral entrapment neuropathy
  Interventions: Drug: 5% dextrose

INTERVENTIONS:
Drug: platelet-rich plasma — Ultrasound-guided 3cc PRP injection between medial epicondyle and ulnar nerve
  Arms: platelet-rich plasma
Drug: 5% dextrose — Ultrasound-guided 3cc 5% dextrose injection between medial epicondyle and ulnar nerve
  Arms: 5% dextrose

SUMMARY:
Ulnar neuropathy at elbow (UNE) is the second common peripheral entrapment neuropathy after carpal tunnel syndrome (CTS). Although many conservative managements of UNE were found, their effectiveness were often unsatisfied without existed guideline. Recently, the perineural injection of 5% dextrose wate (D5W) is a novel management for CTS but its effect for UNE is not obviously as CTS. Hence, it is very important to find another novel injectate for UNE.

DETAILED DESCRIPTION:
The platelet-rich plasma (PRP) is a new and potential treatment for patients with kinds of musculoskeletal disorders and recent reports showed being beneficial for peripheral neuropathy in animal studies. Our previous research shown single injection with PRP was superior to D5W for CTS. However there is no study investigating the effect of PRP for UNE now. Hence, the purpose of this study was to assess the effect of perineural PRP injection for UNE.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20-80 year-old.
2. Diagnosis as ulnar neuropathy at elbow at least one month

Exclusion Criteria:

1. Cancer
2. Coagulopathy
3. Pregnancy

3. Any active infection status 4. Polyneuropathy of upper extremity 5. Brachial plexopathy 6. Thrombocytopenia Previously undergone wrist surgery or steroid injection for ulnar neuropathy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | Change from baseline at 6 month after injection
  Digital pain severity or paresthesia/dysthesia was evaluated using VAS. Pain score scale ranged from 0 to 10, with 10 indicating the most severe pain.

SECONDARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand (DASH) | Change from baseline at 6 month after injection
  Taiwan Disabilities of the Arm, Shoulder and Hand (DASH) contains 11-item disability/symptom scale and each item has five levels of response scoring from 1 to 5. The higher score means more disability or severer symptoms.
Electrophysiological study | Change from baseline at 6 month after injection
  Nerve motor conduction velocity of the ulnar nerve before treatment and multiple time frame after treatment.
Cross-sectional area of ulnar nerve | Change from baseline at 6 month after injection
  Using the musculoskeletal sonogram to measure the cross-sectional area of the ulnar nerve before treatment and multiple time frame after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Tsan Wu, Principal Investigator — Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Locations (1):
- Yung-Tsan Wu, Taipei, Neihu District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Shen YP, Li TY, Chou YC, Ho TY, Ke MJ, Chen LC, Wu YT. Comparison of perineural platelet-rich plasma and dextrose injections for moderate carpal tunnel syndrome: A prospective randomized, single-blind, head-to-head comparative trial. J Tissue Eng Regen Med. 2019 Nov;13(11):2009-2017. doi: 10.1002/term.2950. Epub 2019 Aug 20. PMID 31368191
- [Result] Wu YT, Ke MJ, Ho TY, Li TY, Shen YP, Chen LC. Randomized double-blinded clinical trial of 5% dextrose versus triamcinolone injection for carpal tunnel syndrome patients. Ann Neurol. 2018 Oct;84(4):601-610. doi: 10.1002/ana.25332. Epub 2018 Oct 4. PMID 30187524
- [Result] Wu YT, Ho TY, Chou YC, Ke MJ, Li TY, Huang GS, Chen LC. Six-month efficacy of platelet-rich plasma for carpal tunnel syndrome: A prospective randomized, single-blind controlled trial. Sci Rep. 2017 Dec;7(1):94. doi: 10.1038/s41598-017-00224-6. Epub 2017 Mar 7. PMID 28273894